CLINICAL TRIAL: NCT00817206
Title: Ph3, Open Label, Multi-Ctr, Pros, Rand Study -Efficacy and Safety, Conversion Prograf® Capsules BID to LCPTacro Tablets QD, for Prevent of Acute Allograft Rejection in Stable Kidney Transplant pt.
Brief Title: Safety and Efficacy of LCP-Tacro™ Once Daily in Stable Renal Transplant Patients Converted From Prograf® Twice Daily
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCP-Tacro 3001
Record Dates: First submitted 2008-12-19; First posted 2009-01-06 (Estimated); Results first posted 2015-09-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-08

CONDITIONS: Renal Failure
Keywords: kidney transplantation; renal transplantation; maintenance immunosuppression; tacrolimus; Prevention of acute allograft rejection
MeSH Terms: conditions — Renal Insufficiency | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LCP-Tacro (Experimental): LCP-Tacro tablets™, once daily (LifeCycle Pharma A/S, Hoersholm DK)
  Interventions: Drug: LCP-Tacro
- Prograf (tacrolimus) (Active Comparator): Prograf® capsules, twice daily (Astellas Pharma US, Deerfield IL)
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: LCP-Tacro — LCP-Tacro tablets will be administered orally QD, at the same time in the morning to maintain trough levels at 5-15 ng/ML. Subsequent doses will be adjusted according to whole blood tacrolimus trough levels. LCP-Tarco (tacrolimus) tablets provided in 0.5 mg, 1 mg, 2 mg, and 5 mg tablets.
  Other Names: tacrolimus; tacrolimus modified release
  Arms: LCP-Tacro
Drug: Prograf — Oral prograf doses will be given BID (in the morning and evening), to maintain trough levels of 5- 15 ng/mL. Prograf capsules (tacrolimus) capsules, twice daily oral, provided in 0.5 mg, 1 mg, and 5 mg capsules.
  Other Names: tacrolimus
  Arms: Prograf (tacrolimus)

SUMMARY:
This is 2-armed parallel group, prospective, randomized, open-label, multicenter Phase 3 controlled trial to establish the efficacy and safety of conversion from maintenance immunosuppressive therapy with Prograf® capsules (tacrolimus, Astellas Pharma US, Inc., Deerfield, IL) twice daily to maintenance immunotherapy with LCP Tacro™ tablets (tacrolimus, LifeCycle Pharma A/S, Hoersholm, Denmark) once daily for the prevention of acute allograft rejection in stable adult kidney transplant patients. Patients on a stable dose of Prograf® will be randomly assigned to be converted from Prograf® twice daily to LCP Tacro™ once daily or to remain on maintenance therapy with Prograf® twice daily. Patients entering the study will be treated with assigned study drug and followed for one year for patient survival and the incidence of graft rejection or graft loss.

DETAILED DESCRIPTION:
This is 2-armed parallel group, prospective, randomized, open-label, multicenter Phase 3 controlled trial to establish the efficacy and safety of conversion from maintenance immunosuppressive therapy with Prograf capsules (tacrolimus, Astellas Pharma US, Inc., Deerfield, IL) twice daily to maintenance immunotherapy with LCP-Tacro tablets (tacrolimus, LifeCycle Pharma A/S, Horsholm, Denmark) once daily for the prevention of acute allograft rejection in stable adult make and female kidney transplant patients. Recipients of kidney transplant 3 months to 5 years before Screening and on a stable dose of Prograf will be randomly assigned to be converted from Prograf twice daily to LCP-Tacro once daily or to remain on maintenance therapy with Prograf twice daily. There will be 11 study visits in the Treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years of age who are recipients of a kidney transplant between 3 months and 5 years before the screening date
* Patients taking oral Prograf® capsules twice daily, at least 2 mg total dose per day, as part of their maintenance immunosuppression therapy, with tacrolimus trough levels of 5 to 15 ng/mL
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days before receiving study drug

Exclusion Criteria:

* Recipients of any transplanted organ other than kidney
* Recipients of a bone marrow transplant
* Patients with an eGFR (MDRD7) < 30 mL/min at Screening
* Patients with a spot protein:creatinine ratio > 0.5
* Patients with a WBC count ≤ 2.8 ´ 109/L unless the WBC count has been stable for at least 2 weeks and the absolute neutrophil count is > 1.0 ´ 109 /L
* Patients unable to swallow study medication
* Patients incapable of understanding the purposes and risks of the study, who cannot give written informed consent and who are unwilling or unable to comply with the study protocol requirements
* Pregnant or nursing women
* Patients with reproductive potential who are unwilling/unable to use a double barrier method of contraception
* Patients who were treated with any other investigational agent within 3 months before Screening
* Patients who have taken sirolimus or everolimus within 3 months before Screening
* Patients on concurrent immunosuppression with MMF (CellCept) or MPS delayed-release tablets (Myfortic) who have not been on stable doses for at least 4 weeks before Screening
* Patients withdrawn from corticosteroids less than 30 days before Screening
* Patients with an episode of acute rejection requiring antibody therapy within 3 months before Screening
* Patients treated for acute rejection within 30 days before Screening
* Patients who are hepatitis C virus (HCV) negative who have received an HCV positive (HCV RNA by polymerase chain reaction or HCV antibody) donor kidney
* Patients seropositive for human immunodeficiency virus
* Patients with a current malignancy or a history of malignancy (within the past 5 years), except basal or nonmetastatic squamous cell carcinoma of the skin that has been treated successfully
* Patients with uncontrolled concomitant infection, a systemic infection requiring treatment, or any other unstable medical condition that could interfere with the study objectives
* Patients with severe diarrhea, vomiting, active peptic ulcer, or gastrointestinal disorder that may affect the absorption of tacrolimus
* Patients with any form of current substance abuse, psychiatric disorder, or a condition that, in the opinion of the investigator, may invalidate communication with the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2008-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Steinberg, M.D., Principal Investigator — Claifornia Institute of Renal Research/Sharp Memorial
Locations (1):
- California Institute of Renal Research/ Sharp Memorial, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Started | 163 | 163
Completed | 142 | 154
Not Completed | 21 | 9
Not completed — Adverse Event | 10 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Population: Demographic information is given for all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | LCP-Tacro | Prograf (Tacrolimus) | Total
Number analyzed (Participants) | 163 | 163 | 326
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 146 | 137 | 283
  >=65 years | 17 | 26 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (11.71) | 50.2 (13.49) | 50.3 (1.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 61 | 107
  Male | 117 | 102 | 219
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 29 | 55
  Not Hispanic or Latino | 137 | 134 | 271
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 36 | 34 | 70
  White | 120 | 117 | 237
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 122 | 121 | 243
  Europe | 41 | 42 | 83

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint for Efficacy Failure Within 12 Months of Randomization: Death, Graft Failure, Biopsy-proven Acute Rejection or Loss to Follow-up.
Time Frame: 12 months
Population: One patient in each arm were randomized but not treated. Only treated patients (modified ITT population) is included in the primary outcome measure.
  One patient death is listed under the Prograf arm; this patient died during follow up and did completet the study.
Measure: Number; unit: participants
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Number analyzed (Participants) | 162 | 162
participants
  Death | 2 | 1
  Graft Failure | 0 | 0
  BPAR | 1 | 4
  Loss to follow up | 0 | 1

ADVERSE EVENTS:
Time Frame: SAEs were collected for 1 year for all patients receiving at least one dose of study drug (mITT population).
Arm/Group | LCP-Tacro | Prograf (Tacrolimus)
Serious Adverse Events (participants affected / at risk) | 36/162 | 26/162
Other Adverse Events (participants affected / at risk) | 135/162 | 133/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=162) | Prograf (Tacrolimus) (N=162)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrilation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitits (Infections and infestations) | 2 (2) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2)
Emphysematous pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (3) | 0 (0)
Pneumococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Polyomavirus-associated nephropathy (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (4)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral Pericarditis (Infections and infestations) | 0 (0) | 1 (1)
Vulval cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
Epstein-Barr virus test positive (Investigations) | 1 (1) | 0 (0)
Diabetis mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sqaumous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (2)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax spontaneous tension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arterial disorder (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=162) | Prograf (Tacrolimus) (N=162)
Diarrhoea (Gastrointestinal disorders) | 22 (31) | 15 (17)
Nausea (Gastrointestinal disorders) | 10 (13) | 6 (6)
Nasopharyngitis (Infections and infestations) | 15 (16) | 18 (24)
Urinary tract infection (Infections and infestations) | 14 (19) | 22 (39)
Upper respiratory tract infection (Infections and infestations) | 12 (13) | 14 (16)
Blood creatinine increased (Investigations) | 20 (20) | 14 (16)
Oedema Peripheral (General disorders) | 11 (12) | 10 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (10) | 9 (11)
Headache (Nervous system disorders) | 15 (18) | 11 (12)
Dizziness (Nervous system disorders) | 9 (10) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (8)
Hypertension (Vascular disorders) | 7 (8) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other